CLINICAL TRIAL: NCT04538911
Title: Randomized, Blinded, Single-arm Intradermal Injection, Control of Similar Products on the Market, the Safety Pre-evaluation Phase I Clinical Trial of BCG-PPD in Tuberculosis Patients
Brief Title: Phase I Clinical Protocol for Pre-evaluation of the Safety of BCG-PPD in Tuberculosis Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Shenzhen Third People's Hospital (Other); Beijing Kangterike Statistical Technology Co., Ltd. (Unknown); Wuhan Pulmonary Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: LKM-2020-PPD02
Record Dates: First submitted 2020-08-28; First posted 2020-09-04 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Tuberculosis
Keywords: diagnosis of tuberculosis; epidemiological investigation of tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 30 tuberculosis patient were randomly assigned to the experimental group and the control group. The experimental group was injected with BCG-PPD drug once, while the control group was injected with BCG-PPD drug once
  Interventions: Drug: BCG-PPD
- control group (Other): 30 tuberculosis patient were randomly assigned to the experimental group and the control group. The experimental group was injected with BCG-PPD drug once, while the control group was injected with BCG-PPD drug once
  Interventions: Drug: BCG-PPD

INTERVENTIONS:
Drug: BCG-PPD — BCG-PPD was used for skin test in 30 TB patients, and BCG-PPD was marketed in other 30 TB patients (as control)

SUMMARY:
A total of 60 TB patients aged 65 years and below who are randomly assigned to the experimental group and the control group. The experimental group is injected with BCG-PPD test drug once, and the control group is injected with BCG-PPD control drug once.Subjects undergoing physical examination, vital signs, blood routine, urine routine, blood biochemistry, electrocardiogram, chest X-ray, tuberculosis culture, tuberculosis smear, HIV antibody test and blood pregnancy（only women of childbearing age） during the screening period.Vital signs were checked before skin test, the injection site is photographed at 0min after skin test, and vital signs are checked at 30min after skin test.Vital signs examination, injection site photography and reaction measurement are performed 48h and 72h after skin test.Physical examination, vital signs, routine blood test, routine urine test, biochemical test, electrocardiogram and blood pregnancy test are performed again 7 days after skin test to evaluate the safety of BCG-PPD.

DETAILED DESCRIPTION:
Prior to the commencement of the study, the Investigator/his authorized officer will contact the subject and/or guardian to enroll the candidate subjects and invite them to participate in the study.Subjects who are eligible for screening receive the drug number in the order they arrive at the random number allocation room.They have to undergoing physical examination, vital signs, blood routine, urine routine, blood biochemistry, electrocardiogram, chest X-ray, tuberculosis culture, tuberculosis smear, HIV antibody test and blood pregnancy（only women of childbearing age） during the screening period. Inverstigator absorb and inject 0.1ml drug into the upper and middle 1/3 of the left forearm by Mondo's method. The reaction of the injection site was checked and photographed at 0min, 48h and 72h after the skin test. Meanwhile, the transverse and longitudinal diameers of skin induration and redness were measured at 48h and 72h after the skin test.Vital signs are checked at 30min after skin test.Vital signs examination, injection site photography and reaction measurement are performed 48h and 72h after skin test.Physical examination, vital signs, routine blood test, routine urine test, biochemical test, electrocardiogram and blood pregnancy test are performed again 7 days after skin test.All AE occurred within 7 days after skin test were recorded by a diary card. AE related to the test drug should be followed up to the end of the event.Skin test of subjects aged 18-45 years shall be conducted first. After safety assessment, skin test of subjects aged 46-65 years old, 6-17 years old and under 6 years old shall be conducted successively.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for tuberculosis patients:

  1. Subjects aged 15 ~ 65 years (including 15 and 65 years old) who are clinically diagnosed or diagnosed with tuberculosis.
  2. Subjects under the age of 15 (excluding those under the age of 15) who are clinically diagnosed or diagnosed with tuberculosis.
  3. I (and/or my guardian) agree to participate in the study and sign the informed consent.
  4. I (and/or guardian) can comply with the requirements of the clinical trial protocol to participate in the follow-up.
* Inclusion criteria for patients with extrapulmonary tuberculosis:

  1. The patient was diagnosed with extrapulmonary tuberculosis by epidemiology, clinical manifestations, imaging examination, etiology examination, pathology examination and other auxiliary examinations, and the tuberculosis focus involved other parts of the lung.Combined with the characteristics of this clinical study and field implementation, the inclusion of patients with extrapulmonary tuberculosis should meet the "chemotherapy intensification period not completed".
  2. I (and/or my guardian) agree to participate in the study and sign the informed consent.
  3. I (and/or guardian) can comply with the requirements of the clinical trial protocol to participate in the follow-up.

Exclusion Criteria:

1. Suffering from acute infectious diseases (such as measles, pertussis, influenza, pneumonia, etc.), acute ophthalmic membranitis, acute otitis media, extensive skin diseases and allergic constitution(A history of allergy to two or more drugs or foods, or a known allergy and scar constitution to this drug component).
2. People have any serious disease, such as: tumor, progressive atherosclerosis or diabetes with complications, chronic obstructive pulmonary disease requiring oxygen therapy, acute or progressive liver or kidney disease, congestive heart failure, etc.
3. Convulsion, epilepsy, history of mental illness and/or family history of mental illness.
4. Patients with known or suspected (or high-risk) immune function impairment or abnormality,For example, patients receiving immunosuppressive or immunobooster therapy, patients receiving glucocorticoids, immunoglobulin preparations or blood products or plasma extracts outside the gastrointestinal tract within 3 months, human immunodeficiency virus infection or related diseases.
5. The test results of human immunodeficiency virus (HIV) antibody are positive.
6. Before enrollment, the interval between inoculation of live attenuated vaccine is less than 28 days, and the interval between inoculation of other vaccines is less than 14 days.
7. In the acute stage of disease or acute onset of chronic disease (3 days before skin test).
8. People are participating in or has participated in any other clinical investigator within 3 months prior to this clinical study.
9. Pregnant or lactating women, or planning to become pregnant during the study period.
10. A clear history of hypertension.
11. Suspected or confirmed drug abuse or alcohol abuse.
12. persons with upper limb disabilities.
13. Infants (under one year of age) whose birth weight is less than 2.5kg, or premature or refractory infants.
14. Infants (under 1 year of age) suffering from neonatal respiratory distress syndrome, pathological jaundice, congenital malformations, developmental disorders and congenital diseases.
15. The investigator believes that there are any conditions such as poor compliance that may affect the evaluation of the trial.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence of all adverse event and results of laboratory tests | 7 days after injection
  Record and evaluate the incidence of all adverse event within 7 days after injection；Record and evaluate abnormal incidence of blood routine, urine routine, blood biochemical and electrocardiogram indicators 7 days after injection
Evaluate the effectiveness of the product by measuring the size of the skin response | Between 48 and 72 hours after injection
  The transverse and longitudinal diameters (millimetre) of skin induration and redness, as well as local double circles, blisters, necrosis, and lymphangitis, were recorded at 48h and 72h after injection

CONTACTS AND LOCATIONS:
Overall Officials: Shuihua Lu, Bachelor, Principal Investigator — Shenzhen Third People's Hospital; Hai Huang, Bachelor, Principal Investigator — Wuhan Pulmonary Hospital; Guan Liu, Master, Principal Investigator — Wuhan Pulmonary Hospital
Locations (1):
- The Third People's Hospital Of Shenzhen, Shenzhen, Guangdong, China